CLINICAL TRIAL: NCT06378671
Title: Single-center Clinical Study on the Safety and Effect of Bronchoscopic Cryotherapy in Patients With Chronic Cough
Acronym: ColdCough
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Collaborators: Ningbo SensCure Biotechnology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Li Shiyue, professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ColdCough
Record Dates: First submitted 2024-04-07; First posted 2024-04-22 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Chronic Cough
Keywords: Chronic Cough; Cryotherapy treatment via bronchoscopy
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Intervention Model Description: a prospective, single-center, double-blind ,randomized controlled clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy Treatment (Experimental): The plan is to enroll 20 patients, who will be randomly assigned in a 1:1 ratio to the experimental group and the control group according to the protocol criteria. The experimental group will undergo routine bronchoscopy examination, lavage, and mucosal biopsy, followed by cryotherapy treatment locally (around the left and right main bronchi, upper trachea, and carina).
  Interventions: Procedure: General treatment; Procedure: Cryotherapy Treatment
- Not receiving cryotherapy treatment (Sham Comparator): The plan is to enroll 20 patients, who will be randomly assigned in a 1:1 ratio to the experimental group and the control group according to the protocol criteria. The control group will undergo routine bronchoscopy examination, lavage, and mucosal biopsy.
  Interventions: Procedure: General treatment

INTERVENTIONS:
Procedure: General treatment — routine bronchoscopy examination, lavage, and mucosal biopsy
Procedure: Cryotherapy Treatment — local cryotherapy treatment (around the left and right main bronchi, upper trachea, and carina)
  Arms: Cryotherapy Treatment

SUMMARY:
Chronic cough is one of the most common complaints in respiratory specialty clinics, imposing significant economic burden on patients and severely affecting their quality of life. Currently, the pathogenesis of chronic refractory cough remains incompletely understood, and treatment remains a major challenge in clinical practice. Cryotherapy treatment via bronchoscopy has shown efficacy in certain airway diseases, but there is currently no research reporting its effects on chronic refractory cough.

The goal of this clinical trial is to learn if Cryotherapy treatment works to treat individuals with chronic cough. It will also learn about The safety and effectiveness of the cryotherapy treatment system produced by Ningbo SensCure Biotechnology Co., Ltd.. The main questions it aims to answer are:

* Does cryotherapy treatment lower the frequency and severity of cough and enhance quality of life?
* Will there be safety or operational performance issues when using this cryotherapy treatment system? Researchers will compare cryotherapy treatment with no treatment to determine if cryotherapy treatment is effective for treating chronic cough.

Participants will:

* Take routine bronchoscopy examination, lavage, and mucosal biopsy ,with/without cryotherapy treatment locally (around the left and right main bronchi, upper trachea, and carina)
* undergo a screening period of approximately 28 days. Follow-up visits and necessary examinations will be scheduled for the 3rd day after treatment initiation and at weeks 1, 2, 4, 8, and 12 thereafter.
* Monitor vital signs and clinical manifestations.

DETAILED DESCRIPTION:
1. Objective The objective is to treat patients with chronic cough using the cryotherapy treatment system (including cryotherapy ablation equipment and associated cryotherapy ablation catheters) to improve cough symptoms and enhance patient quality of life. Additionally, to evaluate the safety and effectiveness of the cryotherapy treatment system produced by Ningbo SensCure Biotechnology Co., Ltd., and to provide scientifically reliable data for further formal clinical trials.
2. content This is a prospective, randomized, controlled, small-sample clinical trial, with plans to enroll 20 participants. The experimental device is the cryotherapy treatment system developed and manufactured by Ningbo SensCure Biotechnology Co., Ltd. (including cryotherapy ablation equipment and associated cryotherapy ablation catheters). Safety evaluation criteria (including the incidence of device/procedure-related serious adverse events, device/procedure adverse event rate, incidence of serious adverse events, and device defect rate) and effectiveness evaluation criteria (including cough visual analog scale score, number of coughs within 2 hours, modified cough score scale, Leicester Cough Questionnaire, and cough sensitivity testing) will be used to assess the safety and effectiveness of the cryotherapy treatment system for treating patients with chronic cough.
3. Criteria and Procedures for Withdrawal/Termination of Trial Treatment

Subjects may prematurely terminate treatment or withdraw from the study due to any of the following, but not limited to:

1. Medical or safety reasons deemed necessary by the investigator for the subject to withdraw from the study;
2. Failure to meet inclusion criteria or meeting exclusion criteria after enrollment;
3. Subject's unwillingness to continue participating in the study for any reason;
4. Loss to follow-up (the investigator is unable to contact the subject to return to the clinic for primary endpoint assessment and examination);
5. Termination of the study requested by the investigator or the company for any reason.

For all subjects who prematurely terminate the study, the investigator should obtain the reason for withdrawal as much as possible, such as adverse events, correction of ineffective treatment, withdrawal from the trial based on the investigator's decision, or other reasons, and the withdrawal reason should be recorded in the Case Report Form (CRF).

4．Expected Duration of Participation for Each Subject The expected duration of participation for each subject is defined as the time from the subject's signing of the informed consent form to the end of the final follow-up visit. According to the trial design, the visit schedule for each subject is as follows: Visit 1 (screening period, pre-operative -28 days to treatment period), Visit 2 (treatment period, Day 0), Visit 3 (Day 3 ± 1 day), Visit 4 (Week 1 ± 1 day), Visit 5 (Week 2 ± 3 days), Visit 6 (Week 4 ± 3 days), Visit 7 (Week 8 ± 7 days), and Visit 8 (Week 12 ± 7 days).

5．Monitoring Plan Executor: Monitor. Monitoring Content: Whether the trial protocol is followed; whether all Case Report Form (CRF) entries are correct, complete, and consistent with the original documents such as medical records and physical examination reports, and whether there are any errors or omissions in the data. Since most of the data in the CRF are transcribed from original sources such as medical records and physical examination reports, much of the content is secondary data. Therefore, during monitoring, the content of the CRF needs to be meticulously cross-checked with the original documents to ensure that the data in the CRF are completely consistent with the original data. This process is also known as Source Data Verification (SDV).

6．Data Management and Statistical Analysis Methods A separate data folder will be established for each participant, and dedicated personnel will be responsible for data collection and entry. Adhering to Good Clinical Practice (GCP) principles, it is essential to ensure the authenticity and traceability of the data, retaining all raw data for verification purposes. Statistical analysis of the data will be conducted using SAS 9.4 or higher software.

ELIGIBILITY:
Inclusion Criteria(To be eligible, all of the following criteria must be met):

* Age between 18 and 65 years, regardless of gender;
* Patients with cough of unknown etiology or cause, lasting for more than 8 weeks;
* Cough Visual Analogue Scale (VAS) score ≥ 50；
* Willingness to provide voluntary informed consent and agree to follow-up;
* The investigator believes that the overall status of the subjects does not affect the evaluation and completion of the trial.

Exclusion Criteria(Any one of the following criteria must not be met to be eligible):

* Presence of other diseases that may affect treatment efficacy and prognosis.
* Severe underlying conditions such as heart, brain, or lung diseases.
* Inability to tolerate bronchoscopy procedures and painless anesthesia.
* Women who are pregnant, breastfeeding, or planning pregnancy.
* Intravenous drug users.
* Participation in or currently participating in other clinical studies involving drugs, devices, or other interventions within the month prior to enrollment.
* Other conditions deemed unsuitable for inclusion in this study by the investigators, such as anatomical unsuitability, psychiatric disorders, or psychological disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Device/Surgery-Related Serious Adverse Events | Visit1~Visit8(Preoperative -28 days to week 12±7 days)
  the incidence of device/surgery-related serious adverse events = Number of subjects experiencing device/surgery-related serious adverse events / Total number of subjects receiving cryotherapy treatment × 100%.
Device/Surgery Adverse Event Rate | Visit1~Visit8(Preoperative -28 days to week 12±7 days)
  the incidence rate of device/surgery-related adverse events = Number of subjects experiencing device/surgery-related adverse events / Total number of subjects receiving cryotherapy treatment × 100%.
Serious Adverse Event Rate | Visit1~Visit8(Preoperative -28 days to week 12 ±7 days)
  the incidence rate of serious adverse events = Number of subjects experiencing serious adverse events / Total number of subjects receiving cryotherapy treatment × 100%.
Device Defect Rate | the treatment period(day0)
  the incidence rate of device defects = Number of occurrences of device defects / Total number of times the device was used × 100%.
Cough Visual Analogue Scale (VAS) | during the screening period, the treatment period, day 3, weeks 1, 2, 4, 8, and 12
  Patients will mark on a straight line marked 0-10 cm or 0-100 mm to indicate the severity of cough based on their perception. 0mm(or 0cm) indicates no cough and 100mm(or 10cm) indicates the most severe cough.
Cough frequency within 2 hours | during the screening period and at weeks 4 and 12
  Patients will record the number of coughs they experience within a period of 2 hours based on their perception.
Modified Cough Evaluation Tool (CET) | during the treatment period and at weeks 1, 2, 4, 8, and 12
  The modified CET includes five items assessing patients' daytime cough severity, the impact of nighttime cough on sleep, the intensity of coughing, the impact of coughing on daily life, and its psychological effects. Patients self-assess their coughing based on their experiences over the past week, rating it as "none," "very little," "some," "often," or "frequent."
Leicester Cough Questionnaire (LCQ) | during the treatment period and at weeks 1, 2, 4, 8, and 12
  The Chinese version of the Leicester Cough Questionnaire (LCQ) will be used to assess cough-related quality of life. It consists of 19 questions, which are divided into three health-related dimensions: physiological, psychological and social. Each question is divided into 7 grades, ranging from "All of the time" to "None of the time", according to the degree of severity, with a score ranging from 1 to 7. The score of each dimension is the total score of all the questions in this dimension/the number of questions (score of 1 to 7), and the total score is the sum of the scores of the three dimensions (score of 3 to 21). The higher the score, the better the life and health of patients.
Tracheal Vibratory Cough Stimulation Test | during the screening period and at weeks 4 and 12
  Instruct the subject to look straight ahead. Place the vibrator two fingers above the sternal notch and provide 65Hz vibration stimulation for 10 seconds. Record cough frequency and desire from the start of stimulation to 30 seconds after the end. Coughing or a desire to cough within 30 seconds after the end defines a positive Airway Vibratory Test (AVT).
Capsaicin Cough Stimulation Test | during the screening period and at weeks 4 and 12
  Employ a single-dose inhalation method with a quantified device triggered by inhalation. Begin with saline inhalation as a baseline, followed by incremental inhalation of capsaicin solution at double concentrations (1.95-1000umol/L). Record the number of coughs within 30 seconds after each inhalation.
  Observation indicators: C2, C5 (concentration of capsaicin causing 2 or 5 coughs after inhalation). If coughing doesn't reach 5 times at highest concentration, C5 is considered as 1000μmol/L. The reference value of C5 for this test in normal Chinese individuals is ≥125 μmol/L.
Performance evaluation of Cryotherapy Ablation Equipment | the treatment period(day0)
  Assessed for startup, operational performance, interface user-friendliness, and ease of use. A smooth experiment completion with simple operation is deemed "satisfactory"; otherwise, it's considered "unsatisfactory."
Performance evaluation of Cryotherapy Ablation Catheter | the treatment period(day0)
  Evaluated for operation, cryogenic, and passage performance. Results are categorized as: "satisfactory" for simple operation, successful lesion site arrival, and experiment completion; "fairly satisfactory" for acceptable operation and completion at the lesion site; "fair" for average operation requiring adjustments to reach the lesion site and complete the experiment; "unsatisfactory" for cumbersome operation, failure to reach the lesion site, and experiment failure.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song WJ, Chang YS, Faruqi S, Kim JY, Kang MG, Kim S, Jo EJ, Kim MH, Plevkova J, Park HW, Cho SH, Morice AH. The global epidemiology of chronic cough in adults: a systematic review and meta-analysis. Eur Respir J. 2015 May;45(5):1479-81. doi: 10.1183/09031936.00218714. Epub 2015 Feb 5. No abstract available. PMID 25657027
- [Background] Lai K, Chen R, Lin J, Huang K, Shen H, Kong L, Zhou X, Luo Z, Yang L, Wen F, Zhong N. A prospective, multicenter survey on causes of chronic cough in China. Chest. 2013 Mar;143(3):613-620. doi: 10.1378/chest.12-0441. PMID 23238526
- [Background] Gibson PG, Vertigan AE. Management of chronic refractory cough. BMJ. 2015 Dec 14;351:h5590. doi: 10.1136/bmj.h5590. PMID 26666537
- [Background] Canning BJ, Chang AB, Bolser DC, Smith JA, Mazzone SB, McGarvey L; CHEST Expert Cough Panel. Anatomy and neurophysiology of cough: CHEST Guideline and Expert Panel report. Chest. 2014 Dec;146(6):1633-1648. doi: 10.1378/chest.14-1481. PMID 25188530
- [Background] Nasra J, Belvisi MG. Modulation of sensory nerve function and the cough reflex: understanding disease pathogenesis. Pharmacol Ther. 2009 Dec;124(3):354-75. doi: 10.1016/j.pharmthera.2009.09.006. Epub 2009 Oct 7. PMID 19818366
- [Background] Khalid S, Murdoch R, Newlands A, Smart K, Kelsall A, Holt K, Dockry R, Woodcock A, Smith JA. Transient receptor potential vanilloid 1 (TRPV1) antagonism in patients with refractory chronic cough: a double-blind randomized controlled trial. J Allergy Clin Immunol. 2014 Jul;134(1):56-62. doi: 10.1016/j.jaci.2014.01.038. Epub 2014 Mar 22. PMID 24666696
- [Background] Belvisi MG, Birrell MA, Wortley MA, Maher SA, Satia I, Badri H, Holt K, Round P, McGarvey L, Ford J, Smith JA. XEN-D0501, a Novel Transient Receptor Potential Vanilloid 1 Antagonist, Does Not Reduce Cough in Patients with Refractory Cough. Am J Respir Crit Care Med. 2017 Nov 15;196(10):1255-1263. doi: 10.1164/rccm.201704-0769OC. PMID 28650204
- [Background] Long L, Yao H, Tian J, Luo W, Yu X, Yi F, Chen Q, Xie J, Zhong N, Chung KF, Lai K. Heterogeneity of cough hypersensitivity mediated by TRPV1 and TRPA1 in patients with chronic refractory cough. Respir Res. 2019 Jun 6;20(1):112. doi: 10.1186/s12931-019-1077-z. PMID 31170994
- [Background] Mai Y, Zhan C, Zhang S, Liu J, Liang W, Cai J, Lai K, Zhong N, Chen R. Arnold Nerve Reflex: Vagal Hypersensitivity in Chronic Cough With Various Causes. Chest. 2020 Jul;158(1):264-271. doi: 10.1016/j.chest.2019.11.041. Epub 2020 Jan 13. PMID 31945317
- [Background] Niimi A, Chung KF. Airway inflammation and remodelling changes in patients with chronic cough: do they tell us about the cause of cough? Pulm Pharmacol Ther. 2004;17(6):441-6. doi: 10.1016/j.pupt.2004.09.004. PMID 15564089
- [Background] Niimi A, Torrego A, Nicholson AG, Cosio BG, Oates TB, Chung KF. Nature of airway inflammation and remodeling in chronic cough. J Allergy Clin Immunol. 2005 Sep;116(3):565-70. doi: 10.1016/j.jaci.2005.07.010. PMID 16159625
- [Background] Matsumoto H, Niimi A, Tabuena RP, Takemura M, Ueda T, Yamaguchi M, Matsuoka H, Jinnai M, Chin K, Mishima M. Airway wall thickening in patients with cough variant asthma and nonasthmatic chronic cough. Chest. 2007 Apr;131(4):1042-9. doi: 10.1378/chest.06-1025. PMID 17426208
- [Background] Nakaji H, Niimi A, Matsuoka H, Iwata T, Cui S, Matsumoto H, Ito I, Oguma T, Otsuka K, Takeda T, Inoue H, Tajiri T, Nagasaki T, Kanemitsu Y, Chin K, Mishima M. Airway remodeling associated with cough hypersensitivity as a consequence of persistent cough: An experimental study. Respir Investig. 2016 Nov;54(6):419-427. doi: 10.1016/j.resinv.2016.06.005. Epub 2016 Jul 31. PMID 27886853
- [Background] Hara J, Fujimura M, Ueda A, Myou S, Oribe Y, Ohkura N, Kita T, Yasui M, Kasahara K. Effect of pressure stress applied to the airway on cough-reflex sensitivity in Guinea pigs. Am J Respir Crit Care Med. 2008 Mar 15;177(6):585-92. doi: 10.1164/rccm.200703-457OC. Epub 2008 Jan 10. PMID 18187695
- [Background] Sen RP, Walsh TE. Fiberoptic bronchoscopy for refractory cough. Chest. 1991 Jan;99(1):33-5. doi: 10.1378/chest.99.1.33. PMID 1984981
- [Background] Heching M, Rosengarten D, Shitenberg D, Shtraichman O, Abdel-Rahman N, Unterman A, Kramer MR. Bronchoscopy for Chronic Unexplained Cough: Use of Biopsies and Cultures Increase Diagnostic Yield. J Bronchology Interv Pulmonol. 2020 Jan;27(1):30-35. doi: 10.1097/LBR.0000000000000629. PMID 31651543
- [Background] Sheski FD, Mathur PN. Cryotherapy, electrocautery, and brachytherapy. Clin Chest Med. 1999 Mar;20(1):123-38. doi: 10.1016/s0272-5231(05)70131-3. PMID 10205722
- [Background] Hvidtfeldt M, Pulga A, Hostrup M, Sanden C, Mori M, Bornesund D, Larsen KR, Erjefalt JS, Porsbjerg C. Bronchoscopic mucosal cryobiopsies as a method for studying airway disease. Clin Exp Allergy. 2019 Jan;49(1):27-34. doi: 10.1111/cea.13281. Epub 2018 Oct 12. PMID 30244522
- [Background] Mathur PN, Wolf KM, Busk MF, Briete WM, Datzman M. Fiberoptic bronchoscopic cryotherapy in the management of tracheobronchial obstruction. Chest. 1996 Sep;110(3):718-23. doi: 10.1378/chest.110.3.718. PMID 8797417
- [Background] Zhang L, Yin Y, Zhang J, Zhang H. Removal of foreign bodies in children's airways using flexible bronchoscopic CO2 cryotherapy. Pediatr Pulmonol. 2016 Sep;51(9):943-9. doi: 10.1002/ppul.23361. Epub 2016 Mar 11. PMID 26969845